CLINICAL TRIAL: NCT05659108
Title: iGOGO -Assessment of CPR Skill,Willingness and Public AED in Layperson:A Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200559B0
Record Dates: First submitted 2022-11-16; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Public aid education; cardiopulmonary resuscitation; automated external defibrillators
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CONTROL: stimuli with traditional CPR education per half-year
  Interventions: Behavioral: CPR
- TREATMENT: stimuli with blended CPR education per half-year
  Interventions: Behavioral: CPR

INTERVENTIONS:
Behavioral: CPR — HIGH QUALITY CPR

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is an important public health issue. Chang Gung Memorial Hospital, a university affiliated medical center in Taoyuan city, northern Taiwan, actively cooperated with government policy with 250 automated external defibrillators (AED) donation and implementation around many public places during period of 2012 to 2014. In addition, nearly 200 courses of first aid education and training of citizen were provided in the first and 52 courses in second program. According to the literature, a successful public AED implementation plans proceed with the following requirements: continuing education and training to improve and retain skills; maintaining a proper long-term operation of AED equipment;continued data collection of actual cases for analysis, quality control and feedback. In order to maintain the ability of emergency medical response among these 200 and more AED recipient areas, quality assurance with regular follow-up by medical directors, providing professional advice and feedback, repeat education and training should be proceed.

DETAILED DESCRIPTION:
The aim of study is to continue the research development of the previous projects. First, in the previous research projects, investigators were found that the depth and rate of compression will fall behind the current standards by the American Heart Association after one year of training. The E-learning learning website has been completed, so the new project will launch parallel study and tracking of online (AIR) and field (BASE) stimulation teaching for a 2-year period. The participants would be stimulated at 6 and 18 months with short term on-line or base teaching program, and both groups received tests at 1 and 2 years. Second, NCOV-19 epidemic, many courses were cancelled and cannot be trained normally. Investigators will use feedback Annie to understand the operation status of remote students in online courses, and compare them with traditional field courses. (A1 VS B2) Third, the use of public AED for the first shock in OHCA patients were less than 10% in Taiwan. If the first shock could be saved the time, the prognosis of OHCA patients with shockable rhythm will be greatly improved. Therefore, implementing the early activation of the AED donated by our institute is much important. In the previous simulation test, it was found that the continuous education can activate the public AED 1 minute faster than the unit without training. Therefore, in the new plan, investigators Combined with the pre-hospital rescue data of the Taoyuan Fire Department, investigators will analyse the location of publicAED with the GIS and survival correlation. Fourth, investigators would apply the simulation teaching situation in the hospital to the pre-hospital: try to operate the simulation situation teaching plan of OHCA patients in various public places, so that the students can get the impression of the situation and maintain the skills.

ELIGIBILITY:
Inclusion Criteria:

1. agree to participate in the CPR course and sign the consent form to take part in the trial for further follow-up.
2. satisfies the following age restrictions: a. Legal adult (>20 years old) or b. Underaged (12-20 years old) participants require consent form from the legal guardian.

Exclusion Criteria:

1. Not willing to participate in the trial signed the consent form
2. Inability to perform CPR in a kneeling position
3. unwilling to be tracked
4. Pregnant
5. Hands unable to perform CPR

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recipient of IGOGO AED donation project, other non-profit group and educational institutions, as well as personnel who participated in the initial and recurrent training in the Formosa Plastics Group including Nanya, Formosa Plastics and Chang Gung.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of successful high-quality CPR | we intervention and evaluate the outcome per half-year
  The students stimulate with the traditional education group or blended education per half-year. We evaluate the percentage of successful high-quality CPR between traditional and blended education groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chip-Jin Ng, Dr., Study Chair — Chang Gung Memorial Hospital; Cheng-Yu Chien, Dr., Study Director — Chang Gung Memorial Hospital; Li-Heng Tasi, Dr., Study Director — Chang Gung Memorial Hospital; Ming-Fang Wang, Dr., Principal Investigator — Chang Gung Memorial Hospital; Wei-Chen Chen, Dr., Principal Investigator — Chang Gung Memorial Hospital; Yun-Ting Ku, Researcher, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chien CY, Tsai SL, Huang CH, Wang MF, Lin CC, Chen CB, Tsai LH, Tseng HJ, Huang YB, Ng CJ. Effectiveness of Blended Versus Traditional Refresher Training for Cardiopulmonary Resuscitation: Prospective Observational Study. JMIR Med Educ. 2024 Apr 29;10:e52230. doi: 10.2196/52230. PMID 38683663